CLINICAL TRIAL: NCT02881957
Title: Randomized Clinical Trial of Hypovitaminosis D Treatment in the Neurocritical Care Unit
Brief Title: Hypovitaminosis D in Neurocritical Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Michael Karsy, MD, PhD, MSC, M.D. Ph.D., University of Utah
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB_00091541
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Results first posted 2020-08-17 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-05

CONDITIONS: Craniocerebral Trauma; Intracranial Aneurysm; Brain Neoplasms; Spinal Cord Injuries; Seizures; Meningitis; Stroke; Intracranial Hemorrhages; Critical Illness; Vitamin d Deficiency
Keywords: critical illness; craniocerebral trauma; intracranial aneurysm; spinal cord injuries; seizures; meningitis; stroke; vitamin d deficiency; cholecalciferol; intracranial hemorrhages
MeSH Terms: conditions — Craniocerebral Trauma; Intracranial Aneurysm; Brain Neoplasms; Spinal Cord Injuries; Seizures; Meningitis; Stroke; Intracranial Hemorrhages; Critical Illness; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): Placebo control (simple oral syrup)
  Interventions: Other: Placebo
- Vitamin D3 (Experimental): Cholecalciferol/Vitamin D3 (540,000 IU orally or by feeding tube once)
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol
  Other Names: vitamin D3
  Arms: Vitamin D3
Other: Placebo — Oral syrup placebo
  Arms: Control

SUMMARY:
Vitamin D has been shown to impact prognosis in a variety of retrospective and randomized clinical trials within an intensive care unit (ICU) environment. Despite these findings, there have been no studies examining the impact of hypovitaminosis D in specialized neurocritical care units (NCCU). Given the often significant differences in the management of patients in NCCU and more generalized intensive care units there is a need for further inquiries into the impact of low vitamin D levels in this specific environment. This study proposes a randomized, double-blinded, placebo-controlled, single center evaluation of vitamin D supplementation in the emergent NCCU patient population. The primary outcome will involve length-of-stay for emergent neurocritical care patients. Various secondary outcomes, including in-hospital mortality, ICU length-of-stay, Glasgow Outcome Score on discharge, complications and quality-of-life metrics. Patients will be followed for 6 months post-discharge.

DETAILED DESCRIPTION:
Vitamin D has been shown as an important marker of prognosis in a variety of clinical settings, including overall mortality, acute respiratory distress syndrome (ARDS), infection/sepsis, asthma, cardiovascular disease, diabetes, and pediatric/medical/surgical intensive care unit outcomes. Vitamin D not only plays a role in bone maintenance, but also a variety of extra-axial functions including immune-dysregulation and systemic inflammation. In addition, a number of randomized clinical trials support the supplementation of vitamin D as improving outcome in critical care patients. While the evaluation of vitamin D levels remains a standard-of-care at our institution, the widespread use of vitamin D monitoring and impact on neurocritical care patients remains limited. The investigators' recent prospective observational study of vitamin D levels in neurocritical patients showed that deficiency (<20ng/dL) was highly associated with prolonged hospital stay and increased in-hospital mortality for emergent patients. Moreover, a number of limitations arise from this study due to its observational nature. This study proposes a randomized, double-blinded, placebo-controlled, single center evaluation of vitamin D supplementation in the neurocritical care patient population. Patients admitted to the neurocritical care unit for emergent cases and with vitamin D deficiency (<20ng/dL) will undergo vitamin D serum draw on admission and be randomized to receive cholecalciferol/vitamin D3 supplementation (540,000 IU once orally) or placebo. The primary outcome measured will be hospital length-of-stay. Secondary outcomes will include length of ICU course, complications, medication adverse events, discharge Glasgow Outcome Score, in-hospital and 30-day mortality, as well as quality-of-life. Power analysis estimates 198 patients will be needed for each subgroup to determine a 2 day difference in length-of-stay, and the study plans to recruit 218 patients per treatment arm to account for dropout, which will take approximately 6-9 months to recruit. Interim analysis and safety monitoring will be performed. The investigators hypothesize that vitamin D supplementation may make a significant impact on reducing morbidity and mortality in the neurocritical care population. The possibility of reducing hospital length of stay and mortality from a simple, safe, and cost-effective intervention such as vitamin D supplementation may be a useful adjuvant treatment in the neurocritical care population.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age
* Patients admitted to the neurosurgery or neurology services
* Patients admitted to a critical care unit
* Informed consent
* Expected to stay in the ICU for 48 hours or more
* Vitamin D deficiency (<20ng/mL)

Exclusion Criteria:

* Patients where a vitamin D level was not drawn within 48 hours of admission
* Patients not randomized within 48 hours of admission
* Readmitted patients to the critical care unit
* Lack of informed consent
* Prior supplementation with vitamin D
* Severely impaired gastrointestinal function
* Other trial participation
* Pregnant or lactating women
* Hypercalcemia (total calcium of >10.6 mg/dL or ionized serum calcium of >5.4 mg/dL
* Tuberculosis history or clinical exam
* Sarcoidosis history or clinical exam
* Nephrolithiasis within the prior year
* Patients not deemed suitable for study participation (ie, psychiatric disease, living remotely from the clinic, or prisoner status)
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Karsy, MD, PhD, Principal Investigator — University of Utah, Department of Neurosurgery, Salt Lake City, UT; Min S Park, MD, Study Director — University of Utah, Department of Neurosurgery, Salt Lake City, UT
Locations (1):
- University of Utah Hospital, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guan J, Karsy M, Brock AA, Eli IM, Ledyard HK, Hawryluk GWJ, Park MS. A prospective analysis of hypovitaminosis D and mortality in 400 patients in the neurocritical care setting. J Neurosurg. 2017 Jul;127(1):1-7. doi: 10.3171/2016.4.JNS16169. Epub 2016 Jul 1. PMID 27367248
- [Background] Carter BS, Barker FG. Editorial. Choices in clinical trial design. J Neurosurg. 2019 Sep 13;133(4):1100-1102. doi: 10.3171/2019.7.JNS183276. Print 2020 Oct 1. No abstract available. PMID 31518987
- [Result] Karsy M, Guan J, Eli I, Brock AA, Menacho ST, Park MS. The effect of supplementation of vitamin D in neurocritical care patients: RandomizEd Clinical TrIal oF hYpovitaminosis D (RECTIFY). J Neurosurg. 2019 Sep 13;133(4):1103-1112. doi: 10.3171/2018.11.JNS182713. Print 2020 Oct 1. PMID 31518978
- See also: University of Utah, Department of Neurosurgery — http://medicine.utah.edu/neurosurgery/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo control (simple oral syrup)
  Placebo: Oral syrup placebo
- Vitamin D3: Cholecalciferol/Vitamin D3 (540,000 IU orally or by feeding tube once)
  Cholecalciferol
Period: Overall Study
Arm/Group | Placebo | Vitamin D3
Started | 136 | 138
Completed | 133 | 134
Not Completed | 3 | 4
Not completed — Comfort care | 0 | 1
Not completed — Concurrent trial enrollment | 0 | 1
Not completed — Discharged within 48 hours | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Vitamin D3: Patient demographics of patients receiving study drug
- Placebo: Patient demographics of patients receiving placebo
- Total: Total of all reporting groups
Arm/Group | Vitamin D3 | Placebo | Total
Number analyzed (Participants) | 134 | 133 | 267
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (17.5) | 55.1 (16.8) | 54.0 (17.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 59 | 115
  Male | 78 | 74 | 152
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 15 | 25
  Not Hispanic or Latino | 114 | 102 | 216
  Unknown or Not Reported | 10 | 16 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 5
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Black or African American | 5 | 3 | 8
  White | 107 | 99 | 206
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 18 | 23 | 41
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 134 | 133 | 267

OUTCOME MEASURES:

1. Primary Outcome: Intent-to-treat Hospital Length-of-stay
Description: Intent-to-treat hospital length-of-stay
Time Frame: Until discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 134 | 133
days | 10.9 (15.6) | 9.1 (7.9)
Statistical Analysis 1: Comparison: Vitamin D3 vs Placebo; Two-sided t-test evaluated comparing length of stay in vitamin D3 vs. placebo treated patients utilizing patients as randomized (e.g., intent-to-treat) using a p<0.05 as significant. Adverse events were monitored until discharge; Test type: Superiority; p = 0.2, t-test, 2 sided

2. Primary Outcome: As-treated Hospital Length of Stay
Description: Two-sided t-test evaluated comparing length of stay in vitamin D3 vs. placebo treated patients utilizing patients after randomization, factoring excluded patients (e.g., as-treated) using a p<0.05 as significant.
Time Frame: Until discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 134 | 133
days | 10.4 (14.5) | 9.1 (7.9)
Statistical Analysis 1: Comparison: Vitamin D3 vs Placebo; Test type: Superiority; p = 0.4, t-test, 2 sided

3. Secondary Outcome: Intent-to-treat ICU Length of Stay
Description: Two-sided t-test evaluated comparing length of stay within the ICU specifically in vitamin D3 vs. placebo treated patients utilizing patients after randomization (e.g., intent-to-treat) using a p<0.05 as significant.
Time Frame: Until discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 134 | 133
days | 6.4 (9.8) | 5.4 (6.4)
Statistical Analysis 1: Comparison: Vitamin D3 vs Placebo; Test type: Superiority; p = 0.3, t-test, 2 sided

4. Secondary Outcome: As-treated ICU Length of Stay
Description: Two-sided t-test evaluated comparing length of stay within the ICU specifically in vitamin D3 vs. placebo treated patients utilizing patients after randomization but excluding patients who did not receive treatment (e.g., as-treated) using a p<0.05 as significant.
Time Frame: Until discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 134 | 133
days | 5.8 (7.5) | 5.4 (6.4)
Statistical Analysis 1: Comparison: Vitamin D3 vs Placebo; Test type: Superiority; p = 0.6, t-test, 2 sided

5. Secondary Outcome: In-hospital Mortality
Description: In-hospital mortality
Time Frame: Until discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 134 | 133
Participants | 11 | 13
Statistical Analysis 1: Comparison: Vitamin D3 vs Placebo; Test type: Superiority; p = 0.7, Chi-squared

6. Secondary Outcome: Number of Participants With Study Drug Related Adverse Events
Description: The occurrence of patients who suffered mortality, adverse events or severe adverse events, related specifically to the study drug was monitored. Severe adverse events are defined using common terminology criteria for adverse events (CTCAE) grade 3 or higher specific to vitamin D from time of study drug administration to discharge.
Time Frame: Until discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 134 | 133
Participants | 0 | 0
Statistical Analysis 1: Comparison: Vitamin D3 vs Placebo; Adverse events were monitored until patient discharge from the hospital; Test type: Superiority; p = 0.99, Chi-squared

7. Secondary Outcome: Number of Participants With Sepsis
Description: Diagnosis of sepsis
Time Frame: Until discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 134 | 133
Participants | 2 | 3
Statistical Analysis 1: Comparison: Vitamin D3 vs Placebo; Adverse events were monitored until patient discharge from the hospital; Test type: Superiority; p = 0.6, Chi-squared

8. Secondary Outcome: Number of Participants With Pneumonia
Description: Pneumonia diagnosis
Time Frame: Until discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 134 | 133
Participants | 16 | 14
Statistical Analysis 1: Comparison: Vitamin D3 vs Placebo; Adverse events were monitored until patient discharge from the hospital; Test type: Superiority; p = 0.7, Chi-squared

9. Secondary Outcome: Number of Participants With Urinary Tract Infection
Description: Urinary tract infection diagnosis
Time Frame: Until discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 134 | 133
Participants | 9 | 6
Statistical Analysis 1: Comparison: Vitamin D3 vs Placebo; Adverse events were monitored until patient discharge from the hospital; Test type: Superiority; p = 0.4, Chi-squared

10. Secondary Outcome: Number of Participants With Deep Vein Thrombosis
Description: Deep vein thrombosis diagnosis
Time Frame: Until discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 134 | 133
Participants | 8 | 3
Statistical Analysis 1: Comparison: Vitamin D3 vs Placebo; Adverse events were monitored until patient discharge from the hospital; Test type: Superiority; p = 0.1, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse events were monitored until patient discharge from the hospital.
Description: Catalog of CTCAE grade 3 or 4 adverse events directly related to study drug. Only adverse events or severe adverse events, related specifically to the study drug, were monitored. No serious events in any organ system were identified in this study and thus the listing of only the main heading for Serious Adverse Events and Other (Not Including Serious) Adverse Events reflects this, which is accurate and appropriate.
Arm/Group | Vitamin D3 | Placebo
All-Cause Mortality (participants affected / at risk) | 11/134 | 13/133
Serious Adverse Events (participants affected / at risk) | 0/134 | 0/133
Other Adverse Events (participants affected / at risk) | 0/134 | 0/133

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/57/NCT02881957/Prot_SAP_001.pdf
  • Informed Consent Form (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/57/NCT02881957/ICF_000.pdf